CLINICAL TRIAL: NCT05601999
Title: Multicenter Randomized Single Blind Study of the Clinical Efficacy and Safety of GNR-060 (JSC "GENERIUM", Russia) Compared to Metalyse (Boehringer Ingelheim Pharma GmbH & Co.KG, Germany) in Patients With ST Elevation Myocardial Infarction
Brief Title: Study of Efficacy and Safety of GNR-060 vs Metalyse in Patients With ST Elevation Myocardial Infarction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-STEMI-III; № 142 eff. date 17 March 2021 (Other: Ministry of Health of the Russian Federation)
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Myocardial Infarction; ST Elevation; ECG; STEMI; Myocardial Ischemia; Coronary Thrombosis; Thrombolysis; Thrombolytic; Thrombolytic therapy; Fibrinolytic therapy; Fibrinolysis; Bleeding; Hemorrhagic syndrome; Haemorrhage; Hemorrhagic stroke; Coronary angiography; Revascularization; Reperfusion; Tenecteplase; Metalyse; Metalise; TNK-tPA; Fibrin-specific plasminogen activator; Recombinant DNA technology; AMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Myocardial Ischemia; Coronary Thrombosis; Hemorrhage; Hemorrhagic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNR-060 (Experimental): Main group (122 patients) - GNR-060
  Interventions: Biological: GNR-060
- Metalyse (Active Comparator): Control group (122 patients) - Metalyse
  Interventions: Biological: Metalyse

INTERVENTIONS:
Biological: GNR-060 — GNR-060 will be administered in an individual dose depending on body weight as a single intravenous bolus
  Other Names: Tenecteplase
  Arms: GNR-060
Biological: Metalyse — Metalyse will be administered in an individual dose depending on body weight as a single intravenous bolus
  Other Names: Tenecteplase
  Arms: Metalyse

SUMMARY:
GNR-060(JSC "GENERIUM", Russia) is a proposed biosimilar to the referent product Metalyse. This study is to compare the clinical efficacy and safety of GNR-060 vs Metalyse as a thrombolitic agent in patients with with ST Elevation Myocardial Infarction (STEMI).

DETAILED DESCRIPTION:
The trial is designed as a multicenter randomized single blinded study with the centralized blinded outcome assessment. The patients with diagnosed STEMI will be randomly assigned with one of the treatment options within 4 hours after the symptoms onset. The effectiveness of the tested product GNR-060 or reference product Metalyze will be assessed by the coronarography within 24 hours after the thrombolysis with the following PCI in case of ineffectiveness. The patients will then be followed up for survival and cardiac events for 90 days. The safety assessment will also include any related hemorrhagic complication. The pharmacokinetic parameters and immunogenicity will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction with elevation of the ST segment of the ECG (at point J) in 2 adjacent leads after no more than 6 hours from the onset of pain (lasting at least 20 minutes) in the chest (at the time of screening):

  * ≥ 2.5 mm in male ˂ 40 years, ≥ 2 mm in male ≥ 40 years, or ≥ 1.5 mm in female in leads V2-V3 and/or
  * ≥ 1 mm in other leads in the absence of left ventricular hypertrophy or left bundle branch block.

Exclusion Criteria:

* Diseases accompanied by significant bleeding, currently or within the last 6 months, hemorrhagic diathesis.
* Current oral anticoagulant therapy with INR > 1.3.
* Diseases of the central nervous system at present or in history (neoplasm, aneurysm, surgery on the brain or spinal cord).
* Severe uncontrolled arterial hypertension.
* Major surgical interventions, biopsy of a parenchymal organ or significant trauma within the last 2 months (including trauma in combination with AMI at the present time), recent (within the last 3 months) traumatic brain injury.
* Prolonged or traumatic cardiopulmonary resuscitation (> 2 minutes) within the last 2 weeks.
* Severe liver dysfunction, including liver failure, cirrhosis, portal hypertension (including esophageal varicose veins), active hepatitis.
* Peptic ulcer of the stomach or duodenum in the acute stage.
* Chronic kidney disease or other significant kidney disease with a decrease in glomerular filtration rate ≤30 ml / min / 1.73 m2.
* Arterial aneurysm or presence of arterial/venous vascular malformation.
* Neoplasm with an increased risk of bleeding.
* Acute pericarditis and/or subacute bacterial endocarditis.
* Acute pancreatitis.
* Hypersensitivity to the active substance (tenecteplase), gentamicin (residual traces of the manufacturing process) or any excipient.
* Hemorrhagic stroke or stroke of unknown etiology at present or in history.
* Intracranial (including subarachnoid) hemorrhage at present or in history.
* Ischemic stroke or transient ischemic attack (TIA) within the last 6 months.
* Recent bleeding from the gastrointestinal or genitourinary tract or childbirth (within the last 10 days).
* A recent (before 24 hours) puncture of an incompressible blood vessel (eg, subclavian or jugular vein).
* Congenital and hereditary hemorrhagic coagulopathy (hemophilia, etc.) in history.
* Pregnancy or breastfeeding.
* Body mass index (BMI) less than 18.5 or more than 40 kg/m2.
* Participation in another clinical trial currently or within 30 days prior to screening; use of any investigational drug within 30 days or 5 half-lives prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of the complete myocardial reperfusion based on the independent assessment of coronary angiography | up to 24 hours
  TIMI Grade 3 coronary blood flow after the trombolisis

SECONDARY OUTCOMES:
Frequency of the complete+partial myocardial reperfusion based on the independent assessment of coronary angiography | up to 24 hours
  TIMI Grade 2 or 3 coronary blood flow after the trombolisis
Frequency of myocardial reperfusion based on ECG data | after 90 minutes
  Resolution of the ST segment by 30%, 50%, 70% or more
Changes in troponin T and creatine kinase MB levels | 7 days
90-Day mortality | 90 days
  Mortality within 90 days after myocardial infarction
30-Day and 90-Day cardiovascular mortality | 30 and 90 days
  Cardiovascular mortality up to 30 and 90 days after myocardial infarction
Frequency of the postinfarction complications | up to 30 days
  Frequency of any postifarction complication except for arrythmias
Frequency of the combined events "cardiovascular death + recurrent myocardial infarction + stroke" and "cardiovascular death + recurrent myocardial infarction + stroke + heart failure" | 30 days

OTHER OUTCOMES:
Frequency and severity of hemorrhagic complications | up to 30 days
  Hemorragies will be classified based on BARC, ISTH and TIMI definitions
Incidence of the hemorrhagic stroke | up to 30 days
  Any case of treatment-related hemorrhagic stroke
Frequency and severity of the adverse drug reactions | up to 30 days
  Any adverse events related to the trombolisis
Proportion of patients with the antidrug antibodies | 7 days
  Anti-tenecteplaze antibody will be measured before trombolisis and 7 days after.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, MSc, Study Chair — AO GENERIUM
Locations (11):
- Russia (11):
  - Regional State Budgetary Health Institution "Regional Clinical Emergency Hospital", Barnaul, Altai Territory
  - Regional State Budgetary Institution of Health Care "Altai Territorial Cardiology Dispensary", Barnaul, Altai Territory
  - State Budgetary Institution of Health Care of the Arkhangelsk Region "First City Clinical Hospital named after E.E. Volosevich", Arkhangelsk, Arkhangelskaya oblast
  - Regional State Budgetary Health Institution "Belgorod Regional Clinical Hospital of St. Joasaph", Belgorod, Belgorod Oblast
  - State Autonomous Healthcare Institution of the Perm Territory "City Clinical Hospital No. 4", Perm, Perm Territory
  - Municipal budgetary health care institution "City emergency hospital of the city of Rostov-on-Don", Rostov-on-Don, Rostov Oblast
  - State Budgetary Institution of the Ryazan Region "Regional Clinical Hospital", Ryazan, Ryazan Oblast
  - State budgetary health care institution of the Sverdlovsk region "Scientific and practical center for specialized types of medical care" Ural Institute of Cardiology ", Yekaterinburg, Sverdlovsk Oblast
  - State Autonomous Healthcare Institution "Interregional Clinical and Diagnostic Center", Kazan', Tatarstan Republic
  - State Health Institution "City Clinical Emergency Hospital No. 25", Volgograd, Volgograd Oblast
  - State Budgetary Health Institution of the Yaroslavl Region "Regional Clinical Hospital", Yaroslavl, Yaroslavl Oblast

IPD SHARING:
Plan to Share IPD: No